CLINICAL TRIAL: NCT04468659
Title: AHEAD 3-45 Study: A Placebo-Controlled, Double-Blind, Parallel-Treatment Arm, 216 Week Study With an Extension Phase to Evaluate Efficacy and Safety of Treatment With BAN2401 in Subjects With Preclinical Alzheimer's Disease and Elevated Amyloid (A45 Trial) and in Subjects With Early Preclinical Alzheimer's Disease and Intermediate Amyloid (A3 Trial)
Brief Title: AHEAD 3-45 Study: A Study to Evaluate Efficacy and Safety of Treatment With Lecanemab in Participants With Preclinical Alzheimer's Disease and Elevated Amyloid and Also in Participants With Early Preclinical Alzheimer's Disease and Intermediate Amyloid
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Alzheimer's Clinical Trials Consortium (Other); Biogen (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAN2401-G000-303; R01AG054029 (NIH); R01AG061848 (NIH); 2020-004244-28 (EudraCT Number)
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Preclinical Alzheimer's Disease; Early Preclinical Alzheimer's Disease
Keywords: BAN2401; Preclinical Alzheimer's disease; Elevated amyloid; Early preclinical Alzheimer's disease; Intermediate amyloid; A45 Trial; A3 Trial; AHEAD 3-45; Lecanemab
MeSH Terms: interventions — lecanemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- A45 Trial: Lecanemab 5 mg/kg + 10 mg/kg (Core Study) (Experimental): Participants will receive lecanemab 5 milligram per kilogram (mg/kg), administered as intravenous (IV) infusion, every two weeks from Week 0 to 6, then 10 mg/kg, administered as IV infusion, every two weeks from Week 8 to 94, and 10 mg/kg, administered as IV infusion, every four weeks from Week 96 to 216 in core study.
  Interventions: Drug: Lecanemab
- A45 Trial: Placebo (Core Study) (Placebo Comparator): Participants will receive placebo (0.9 percent [%] sodium chloride solution), administered as IV infusion, every two weeks from Week 0 to 94, then every four weeks from Week 96 to 216.
  Interventions: Drug: Placebo
- A3 Trial: Lecanemab 5 mg/kg + 10 mg/kg (Core Study) (Experimental): Participants will receive lecanemab 5 mg/kg, administered as IV infusion, every four weeks from Week 0 to 4, then 10 mg/kg, administered as IV infusion, every four weeks from Week 8 to 216 in core study.
  Interventions: Drug: Lecanemab
- A3 Trial: Placebo (Core Study) (Placebo Comparator): Participants will receive placebo (0.9% sodium chloride solution), administered as IV infusion, every four weeks from Week 0 to 216.
  Interventions: Drug: Placebo
- A3 and A45 Trial: Lecanemab 10 mg/kg (Extension Phase) (Experimental): Participants (from either A3 or A45 Trial) progressing to early Alzheimer's disease (EAD) during the core study (progressors) will receive lecanemab 10 mg/kg, administered as IV infusion, every two weeks after transition to the extension phase for at least 216 weeks from randomization in the core study. Participants completing the core study (completers) will enter extension phase and will receive lecanemab 5 mg/kg for initial 4 doses, than 10 mg/kg, administered as IV infusion, every two weeks for up to 96 weeks in extension phase.
  Interventions: Drug: Lecanemab

INTERVENTIONS:
Drug: Lecanemab — IV infusion.
  Other Names: BAN2401
  Arms: A3 Trial: Lecanemab 5 mg/kg + 10 mg/kg (Core Study); A3 and A45 Trial: Lecanemab 10 mg/kg (Extension Phase); A45 Trial: Lecanemab 5 mg/kg + 10 mg/kg (Core Study)
Drug: Placebo — IV infusion.
  Arms: A3 Trial: Placebo (Core Study); A45 Trial: Placebo (Core Study)

SUMMARY:
The primary purpose of this study is to determine whether treatment with lecanemab is superior to placebo on change from baseline of the Preclinical Alzheimer Cognitive Composite 5 (PACC5) at 216 weeks of treatment (A45 Trial) and to determine whether treatment with lecanemab is superior to placebo in reducing brain amyloid accumulation as measured by amyloid positron emission tomography (PET) at 216 weeks of treatment (A3 Trial). This study will also evaluate the long-term safety and tolerability of lecanemab in participants enrolled in the Extension Phase.

ELIGIBILITY:
Inclusion criteria:

Participants must meet all of the following criteria to be included in this study:

1. Male or female, age 55 to 80 years inclusive at the time of informed consent, with a plasma biomarker result that is predictive of intermediate or elevated brain amyloid at Screening or known before Screening to have elevated or intermediate amyloid according to previous PET, cerebrospinal fluid (CSF), or plasma testing

   • Those 55 to 64 must have 1 of the following additional risk factors, given the relatively low rates of amyloid positivity less than (<) 65 years, before screening:
   * First degree relative diagnosed with dementia onset before age 75, or
   * Known to possess at least 1 apolipoprotein E4 variant (APOE4) allele, or
   * Known before screening to have elevated brain amyloid according to previous plasma biomarker results, PET imaging, or CSF testing
2. Global Clinical Dementia Rating (CDR) score of 0 at screening
3. Mini Mental State Examination score greater than or equal to (>=) 27 (with educational adjustments) at screening.
4. Wechsler Memory Scale-Revised Logical Memory subscale II (WMS-R LM II) score at screening of >=6
5. A45 Trial: Elevated brain amyloid pathology by amyloid PET: defined as approximately greater than (>) 40 Centiloids on screening scan A3 Trial: Intermediate levels of brain amyloid pathology by amyloid PET: defined as approximately 20 to 40 Centiloids on screening scan
6. Has a study partner that is willing to participate as a source of information and has approximately weekly contact with the participant (contact can be in-person, via telephone or electronic communication). The study partner must have sufficient contact such that the investigator feels the study partner can provide meaningful information about the participant's daily function
7. Provide written (or electronic, if allowed per country-specific regulations) informed consent
8. Willing and able to comply with all aspects of the protocol

For extension phase :

1. Completed the Core Study, or meet the following progression criteria during the Core Study:

   * Two consecutive CDR visits with Global Scores > zero when measured at least 6 months apart within the Core Study
   * The principal investigator's confirmation that the participant has clinically declined consistent progression to EAD
2. Must continue to have a study partner who is willing and able to provide follow-up information on the participant throughout the course of the Extension Phase. The study partner must provide separate written informed consent for the Extension Phase. Study partners must continue to have sufficient contact such that the investigator feels the study partner can provide meaningful information about the participant's daily functions
3. Provide written informed consent for the Extension Phase. If a participant lacks capacity to consent in the investigator's opinion, the participant's assent should be obtained, if required and in accordance with local laws, regulations, and customs, plus the written informed consent of a legal representative (capacity to consent and the definition of a legal representative should be determined in accordance with applicable local laws and regulations). In countries where local laws, regulations, and customs do not permit participants who lack capacity to consent to participate in this study (example, Spain), they will not be enrolled
4. Willing and able to comply with all aspects of the protocol

Exclusion criteria:

Participants who meet any of the following criteria will be excluded from this study:

1. Females who are breastfeeding or pregnant at screening or baseline
2. Females of childbearing potential who:

   • Within 28 days before study entry, did not use a highly effective method of contraception For sites outside of Europe, it is permissible that if a highly effective method of contraception is not appropriate or acceptable to the participant, then the participant must agree to use a medically acceptable method of contraception
3. History of transient ischemic attacks (TIA), stroke, or seizures within 12 months of screening
4. Current or history within the past 2 years of psychiatric diagnosis or symptoms that, in the opinion of the investigator, could interfere with study procedures
5. Contraindications to 3 Tesla magnetic resonance imaging (MRI) scanning, including cardiac pacemaker/defibrillator, ferromagnetic metal implants (example, in-skull and cardiac devices other than those approved as safe for use in MRI scanners), or exhibit other significant pathological findings on brain MRI at Screening
6. Hypersensitivity to any monoclonal antibody treatment
7. Any immunological disease which is not adequately controlled, or which requires treatment with immunoglobulins, systemic monoclonal antibodies (or derivatives of monoclonal antibodies), systemic immunosuppressants, or plasmapheresis during the study
8. Bleeding disorder that is not under adequate control (including a platelet count <50,000 or international normalized ratio [INR] >1.5) at screening
9. Results of laboratory tests conducted during screening that are outside the following limits:

   * Thyroid stimulating hormone (TSH) above normal range
   * Abnormally low (below lower limit of normal [LLN]) serum vitamin B12 levels for the testing laboratory (if participant is taking vitamin B12 injections, level should be at or above the LLN for the testing laboratory). A low vitamin B12 is exclusionary, unless the required follow-up labs (homocysteine and methylmalonic acid [MMA]) indicate that it is not physiologically significant
10. Known to be human immunodeficiency virus (HIV) positive
11. Any other clinically significant abnormalities that in the opinion of the investigator require further investigation or treatment or may interfere with study procedures or safety
12. Malignant neoplasms within 3 years of screening (except for basal or squamous cell carcinoma in situ of the skin, or localized prostate cancer in male participants with treatment cycles completed at least 6 months before screening). Participants who had malignant neoplasms but who have had at least 3 years of documented uninterrupted remission before screening need not be excluded
13. Answer "yes" to Columbia-Suicide Severity Rating Scale (C-SSRS) suicidal ideation Type 4 or 5, or any suicidal behavior assessment within 6 months before screening, at screening, or at baseline, or has been hospitalized or treated for suicidal behavior in the past 5 years before screening
14. Known or suspected history of drug or alcohol abuse or dependence within 2 years before screening or a positive urine drug test at screening. Participants who test positive for benzodiazepines, opioids, or tetrahydrocannabinol (THC) in urine drug testing need not be excluded unless in the clinical opinion of the investigator this is due to potential drug abuse
15. Taking prohibited medications
16. Participation in a clinical study involving:

    * Any anti-amyloid plaque lowering immunotherapy (example, therapeutic monoclonal antibody or active anti-amyloid vaccine) at any time, unless it can be documented that the participant was randomized to placebo or never received study drug
    * Any immunoglobulin therapy, or vaccine within 6 months before Screening, unless it can be documented that the participant was randomized to placebo or never received study drug
    * Lecanemab
    * Any new chemical entities or investigational drug for AD within 6 months before randomization unless it can be documented that the participant received only placebo
    * Any other investigational medication or device study in the 8 weeks or 5 half-lives (whichever is longer) of the medication before randomization unless it can be documented that the participant was in a placebo treatment arm
17. Planned surgery during the pre-randomization phase or within 3 months of randomization, which requires general anesthesia

For extension phase:

1. Discontinued from the Core Study or from study treatment
2. Under study drug interruption due to ARIA or other AE at the time of transition to the extension phase

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2028-12-21 (Estimated); Study Completion 2031-01-16 (Estimated)

PRIMARY OUTCOMES:
A45 Trial: Change From Baseline in Preclinical Alzheimer Cognitive Composite 5 (PACC5) Score at Week 216 | Baseline, Week 216
  PACC5(5 components):Free/cued selective reminding test:number of words recalled without cuing/with cuing(0[worst]-96[best recall]);Delayed Paragraph Recall test: recall of 1 short story(25 bits information),immediately after reading and again after delay of 30 minutes (0[worst]-25[best recall]);Digit-symbol substitution test: Participant uses a key to fill in blank squares as fast as possible in 90 seconds(0[none]-91[best performance]);Mini Mental State Score:to evaluate orientation,memory,attention,concentration,naming,repetition,comprehension and ability to create sentence,to copy 2 overlapping pentagons, scored as number of correctly completed items(0[worse]-30[perfect performance]);Category fluency task: participants generate words in 60 second belonging to a semantic category(total score:number of appropriate words generated per task, higher values indicate better performance).
A3 Trial: Change From Baseline in Amyloid Positron Emission Tomography (PET) Standard Uptake Value Ratio (SUVr) at Week 216 | Baseline, Week 216

SECONDARY OUTCOMES:
A45 Trial: Change From Baseline in Amyloid Positron Emission Tomography (PET) Standard Uptake Value Ratio (SUVr) at Weeks 96 and 216 | Baseline, Week 96, Week 216
A45 Trial: Change From Baseline in tau Positron Emission Tomography (PET) Standard Uptake Value Ratio (SUVr) at Weeks 96 and 216 | Baseline, Week 96, Week 216
A45 Trial: Change From Baseline in Cognitive Function Index (CFI) at Week 216 | Baseline, Week 216
  CFI assessment to assess the participant's perceived ability to perform high-level functional tasks in daily life and sense of overall cognitive functional ability. Study participants (18 questions) and their study partners (15 questions) independently rate the participant's abilities. Total score combines participant and study partner scores, with higher scores indicating greater impairment.
A3 Trial: Change From Baseline in tau Positron Emission Tomography (PET) Standard Uptake Value Ratio (SUVr) at Week 216 | Baseline, Week 216

CONTACTS AND LOCATIONS:
Locations (108):
- United States (73):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - UCI MIND, Irvine, California
  - University of Southern California, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford University, Palo Alto, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Univeristy of California, San Francisco, San Francisco, California
  - University of California, Davis, Walnut Creek, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Advanced Clinical Research Network, Corp, Coral Gables, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - K2 Medical Research - The Villages, Lady Lake, Florida
  - K2 Medical Research, Llc, Maitland, Florida
  - K2 Medical Research, Maitland, Florida
  - Gonzalez MD & Aswad MD Health Sciences, Miami, Florida
  - Wien Center for Clinical Research, Miami Beach, Florida
  - Renstar Medical Research, Ocala, Florida
  - Synexus Clinical Research, Orlando, Florida
  - University of South Florida - Health Byrd Alzheimer Institute, Tampa, Florida
  - Synexus Clinical Research, The Villages, Florida
  - Alzheimer's Research and Treatment Center, Wellington, Florida
  - Charter Research, Winter Park, Florida
  - Emory University, Atlanta, Georgia
  - Columbus Memory Center, PC, Columbus, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas, Fairway, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - Brigham and Woman's Hospital Center for Alzheimer Research and Treatment, Boston, Massachusetts
  - Donald S.Marks, M.D.,P.C., Plymouth, Massachusetts
  - University of Michigan (UMICH), Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - Duke Health Center, Durham, North Carolina
  - AMC Research, Matthews, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University/University Hospitals, Beachwood, Ohio
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Central States Research, LLC, Tulsa, Oklahoma
  - Summit Research Network, Oregon, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital Memory and Aging Program, Providence, Rhode Island
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas, Southwestern MC at Dallas, Dallas, Texas
  - University of North Texas Health Sciences Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
  - National Clinical Research, Inc, Richmond, Virginia
  - University of Washington Memory and Brain Wellness Center, Seattle, Washington
  - SIBCR, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Australia (6):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - CALHN Memory Trials, Adelaide, South Australia
  - Austin Hospital - Medical and Cognitive Research Unit, Ivanhoe, Victoria
  - Alzheimer's Research Australia, Nedlands, Western Australia
- Canada (6):
  - Centricity Research, Hailfax, Nova Scotia
  - True North Clinical Research Inc., New Minas, Nova Scotia
  - True North Clinical Research, New Minas, Nova Scotia
  - Parkwood Institute Main Building, London, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- Japan (13):
  - National Center for Geriatrics and Gerontology, Obu-shi, Aichi-ken
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Kobe University Hospital, Kobe, Hyōgo
  - Shonan Kamakura General Hospital, Kamakura-shi, Kanagawa
  - Koseikai Takeda Hospital, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Medical Corporation Heishinkai OPHAC Hospital, Osaka, Osaka
  - Medical Corporation Heishinkai OPHAC Hospital, Suita-shi, Osaka
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - P-One Clinic, Keikokai Medical Corporation, Hachioji -shi, Tokyo
  - Tokyo Metropolitan Geriatric Hospital, Itabashi-ku, Tokyo
  - National Center of Neurology and Psychiatry, Kodaira-shi, Tokyo
  - ICR Clinical Research Hospital Tokyo, Shinjuku-Ku, Tokyo
- National University Hospital, Singapore, Singapore
- Spain (5):
  - Barcelona Beta Brain Research Center, Barcelona
  - Fundació ACE, Barcelona
  - Fundacion CITA ALZHEIMER, Donostia / San Sebastian
  - Hospital Universitario Quirón Salud Madrid, Madrid
  - Hospital Universitario Marqués de Valdeciila, Santander
- United Kingdom (4):
  - Bristol Brain Centre, Bristol
  - Glasgow Memory Clinic, Glasgow
  - St Pancras Clinical Research, London
  - Imperial Memory Unit, London

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Devanarayan V, Doherty T, Charil A, Sachdev P, Ye Y, Murali LK, Llano DA, Zhou J, Reyderman L, Hampel H, Kramer LD, Dhadda S, Irizarry MC. Plasma pTau217 predicts continuous brain amyloid levels in preclinical and early Alzheimer's disease. Alzheimers Dement. 2024 Aug;20(8):5617-5628. doi: 10.1002/alz.14073. Epub 2024 Jun 28. PMID 38940656
- [Derived] Molina-Henry DP, Raman R, Liu A, Langford O, Johnson K, Shum LK, Glover CM, Dhadda S, Irizarry M, Jimenez-Maggiora G, Braunstein JB, Yarasheski K, Venkatesh V, West T, Verghese PB, Rissman RA, Aisen P, Grill JD, Sperling RA. Racial and ethnic differences in plasma biomarker eligibility for a preclinical Alzheimer's disease trial. Alzheimers Dement. 2024 Jun;20(6):3827-3838. doi: 10.1002/alz.13803. Epub 2024 Apr 17. PMID 38629508
- [Derived] Rissman RA, Langford O, Raman R, Donohue MC, Abdel-Latif S, Meyer MR, Wente-Roth T, Kirmess KM, Ngolab J, Winston CN, Jimenez-Maggiora G, Rafii MS, Sachdev P, West T, Yarasheski KE, Braunstein JB, Irizarry M, Johnson KA, Aisen PS, Sperling RA; AHEAD 3-45 Study team. Plasma Abeta42/Abeta40 and phospho-tau217 concentration ratios increase the accuracy of amyloid PET classification in preclinical Alzheimer's disease. Alzheimers Dement. 2024 Feb;20(2):1214-1224. doi: 10.1002/alz.13542. Epub 2023 Nov 6. PMID 37932961
- [Derived] Kirn DR, Grill JD, Aisen P, Ernstrom K, Gale S, Heidebrink J, Jicha G, Jimenez-Maggiora G, Johnson L, Peskind E, McCann K, Shaffer E, Sultzer D, Wang S, Sperling R, Raman R. Centralizing prescreening data collection to inform data-driven approaches to clinical trial recruitment. Alzheimers Res Ther. 2023 May 2;15(1):88. doi: 10.1186/s13195-023-01235-4. PMID 37131229